CLINICAL TRIAL: NCT01717859
Title: Musculoskeletal Ultrasound in Predicting Early Dose Titration With Tocilizumab
Acronym: RASTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Veena Ranganath, M.D., M.S., Assistant Clinical Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ML28542; ML28542 (Other: Genentech Inc.)
Record Dates: First submitted 2012-10-19; First posted 2012-10-31 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tocilizumab (Other): All subjects will receive tocilizumab.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — All subjects will start at 4mg/kg. After 3 months, if DAS28 > 3.2, dosage will be escalated to 8 mg/kg.
  Other Names: Actemra

SUMMARY:
The purpose of this research study is to determine if a change in inflammation or baseline inflammation seen on the ultrasound is a good indicator of how rheumatoid arthritis patients respond to TCZ 4mg/kg and whether early prediction of dose escalation is possible by utilizing ultrasound inflammatory measures.

DETAILED DESCRIPTION:
This is a 24-week, double blind open label clinical trial study to evaluate 57 active Rheumatoid Arthritis (RA) patients who have moderate to severe disease activity with total Power Doppler Ultrasound (PDUS) >10 of 34 joints evaluated by Ultrasound (US) (at screening to enter into the study). All patients will begin treatment with tocilizumab at a dose of 4mg/kg. Two study sites will recruit patients (UCLA and UF) using the same protocol, after standardizing US acquisition methods, as well as scoring. US synovitis scores will be acquired at screening, baseline, and pre-infusion at 4, 12, 16, and 24 weeks, to be able to determine whether change in pre-infusion synovitis score at 4 weeks can be used to predict change in disease activity at 12 weeks. This will provide evidence to whether such reading is useful in predicting which patients may require escalation of dose from 4 to 8 mg/kg. At 12 weeks, patients not meeting low disease activity within the 4mg/kg (disease activity score DAS28/ Erythrocyte Sedimentation Rate (ESR)-4item<3.2) will increase the tocilizumab dose to 8mg/kg (maximum dose 800mg) in a blinded manner to enable evaluation of these US-focused objectives in the context of the current FDA-approved label. The ultrasound scorer will not know information about patient's disease activity (Tender Joint Count (TJC), Swollen Joint Count (SJC), labs etc) or if there was dose escalation at 12 weeks. The clinical assessor of disease activity will be blinded to the ultrasound scores. Additionally, the patient will also be blinded to dose escalation. If patients in the 4mg/kg arm achieve DAS28<3.2 at 12 weeks, patients will continue with their current dose for the duration of the study. Please see the below Table for details on the blinding plan.

ELIGIBILITY:
Inclusion Criteria

Patients must have rheumatoid arthritis. Patients will be included in the trial based on the following criteria:

1. Patient must meet 1987 American College of Rheumatology (ACR) criteria,
2. Age > 18 years of age,
3. Baseline DAS28/ESR>4.4,
4. Stable concomitant DMARDs for more than 1 month (methotrexate, leflunomide, plaquenil, sulfasalazine, or no DMARDs). However, if the patient is not on DMARD, history of DMARD use required.

   1. If not on DMARD (and the patient satisfies the above statement), the patient can opt for monotherapy with tocilizumab or combination therapy OR
   2. If on biologic monotherapy, can opt for monotherapy with tocilizumab or DMARD combination therapy (ie. patients cannot be on biologic with TCZ)

6) Power Doppler score of >10 at screening.

General Medical Concerns:

* Normal organ function, except if abnormal due to the disease under investigation
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.
* Subject has provided written informed consent.

Exclusion Criteria

A patient will be excluded if the answer to any of the following statements is "yes".

General:

1. Major surgery (including joint surgery) within 8 weeks prior to baseline or planned major surgery within 6 months after baseline.

   Excluded Previous or Concomitant Therapy:
2. Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of baseline.
3. Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies, some examples are CAMPATH, anti-CD4, anti-CD5, anti-CD3.
4. Previous treatment with anti-CD19 and anti-CD20 within 6 months of start of the study.
5. Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline.
6. Immunization with a live/attenuated vaccine within 4 weeks prior to baseline.
7. Previous treatment with TCZ.
8. Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation.
9. Use of prednisone > 10mg at baseline.

   Exclusions for General Safety:
10. History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
11. Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, ulcerative colitis, or Crohn's disease.)
12. Current liver disease as determined by principal investigator unless related to primary disease under investigation
13. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds).
14. Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of baseline or oral antibiotics within 2 weeks prior to baseline.
15. Active Tuberculosis (TB) requiring treatment within the previous 3 years. Patients should be screened for latent TB and, if positive, treated following local practice guidelines prior to initiating TCZ. Patients treated for tuberculosis with no recurrence in 3 years are permitted.
16. Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation.
17. Evidence of active malignant disease, malignancies diagnosed within the previous 5 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured), or breast cancer diagnosed within the previous 5 years.
18. Pregnant women or nursing (breast feeding) mothers.
19. Patients with reproductive potential not willing to use an effective method of contraception.
20. History of alcohol, drug or chemical abuse within 1 year prior to screening.
21. Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation.
22. Patients with lack of peripheral venous access.
23. Body weight of > 150 kg.

    Laboratory Exclusion criteria (at screening):
24. Serum creatinine > 1.6 mg/dL (141 µmol/L) in female patients and > 1.9 mg/dL (168 µmol/L) in male patients. Patients with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rates (GFR) are >30.
25. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN)
26. Total Bilirubin > ULN
27. Platelet count < 100 x 109/L (100,000/mm3)
28. Hemoglobin < 85 g/L (8.5 g/dL; 5.3 mmol/L)
29. White Blood Cells < 3.0 x 109/L (3000/mm3)
30. Absolute Neutrophil Count < 2.0 x 109/L (2000/mm3)
31. Absolute Lymphocyte Count < 0.5 x 109/L (500/mm3)
32. Positive Hepatitis BsAg, or Hepatitis C antibody
33. HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veena Ranganath, MD, MS, Principal Investigator — UCLA David Geffen School of Medicine, Division of Rheumatology
Locations (1):
- UCLA David Geffen School of Medicine, Division of Rheumatology, Los Angeles, California, United States

REFERENCES:
- [Derived] Charles-Schoeman C, Wang J, Shahbazian A, Wilhalme H, Brook J, Kaeley GS, Oganesian B, Ben-Artzi A, Elashoff DA, Ranganath VK. Power doppler ultrasound signal predicts abnormal HDL function in patients with rheumatoid arthritis. Rheumatol Int. 2023 Jun;43(6):1041-1053. doi: 10.1007/s00296-023-05285-7. Epub 2023 Feb 24. PMID 36828925
- [Derived] Morris NT, Brook J, Ben-Artzi A, Martin W, Kermani TA, Avedikian-Tatosyan L, Karpouzas G, Nagam H, Navarro G, Choi S, Taylor MB, Elashoff D, Kaeley GS, Ranganath VK. Doppler ultrasound impacts response to intravenous tocilizumab in rheumatoid arthritis patients. Clin Rheumatol. 2021 Dec;40(12):5055-5065. doi: 10.1007/s10067-021-05857-7. Epub 2021 Jul 16. PMID 34269927
- [Derived] Kuo D, Morris NT, Kaeley GS, Ben-Artzi A, Brook J, Elashoff DA, Ranganath VK. Sentinel joint scoring in rheumatoid arthritis: an individualized power Doppler assessment strategy. Clin Rheumatol. 2021 Mar;40(3):1077-1084. doi: 10.1007/s10067-020-05340-9. Epub 2020 Aug 15. PMID 32803573
- [Derived] Choate EA, Kaeley GS, Brook J, Altman RD, FitzGerald JD, Floegel-Shetty AR, Elashoff DA, Ranganath VK. Ultrasound detects synovitis in replaced and other surgically operated joints in rheumatoid arthritis patients. BMC Rheumatol. 2020 Feb 3;4:8. doi: 10.1186/s41927-019-0107-2. eCollection 2020. PMID 32025629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited through printed and internet advertisements, direct recruitment of study participants, referrals, review of medical records to identify potential participants, and through IRB approved screening protocol and IRB approved study. Patients were recruited starting on 9/24/14. The recruitment continued through November of 2016.
Pre-assignment Details: 16 did not pass inclusion criteria, these patients were not able to be assigned to a study arm: 8 had PDUS<10 4 lab values outside limits
  1. pregnant
  2. changed their mind
  1 was taking prednisone.
  Also:
  4 other patients were assigned to the study arm but were deleted from the study due to the considerations mentioned in the protocol
Period: Overall Study
Arm/Group | Tocilizumab
Started | 54
3 Month | 50
Completed | 44
Not Completed | 10
Not completed — Adverse Event | 5
Not completed — Moved out of state | 1
Not completed — Patient concerned about mental health | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tocilizumab
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.87 (15.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 9
  White | 34
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54
Disease duration [Mean (Standard Deviation); unit: years] | 9.94 (7.50)
Disease Activity Score All Joints (DAS28)/ Erythrocyte Sedimentation Rate (ESR) [Mean (Standard Deviation); unit: units on a scale] — DAS28 is a measure of disease activity in rheumatoid arthritis (RA). DAS stands for 'disease activity score' and the number 28 refers to the 28 joints that are examined in this assessment. The calculation takes into account the number of swollen joints, the number of tender joints (both out of 28 assessed joints), the erythrocyte sedimentation rate (ESR), and a self-reported global assessment of health from the patient. DAS28 ranges from 0 to a maximum of 9.48. A DAS28 more than 5.1 implies active disease, less than 3.2 implies low disease activity, and less than 2.6 implies remission.
  units on a scale | 6.30 (1.03)
Clinical Disease Activity Index (CDAI) [Mean (Standard Deviation); unit: units on a scale] — CDAI stands for "Clinical Disease Activity Index" and is a measure used to assess rheumatoid arthritis activity. This scale sums the count of swollen joints, the count of tender joints (both out of 28 assessed joints), and the final scores of both a patient global health assessment and a care provider global health assessment for the patient on a continuous scale from 0-10. CDAI ranges from 0 to 76, and <2.8 implies remission, <10.0 implies low disease activity, <22.0 implies moderate disease activity, and >22.0 implies high disease activity.
  units on a scale | 39.04 (11.90)
Health Assessment Questionnaire- Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — HAQ-DI stands for Health Assessment Questionnaire- Disability Index. HAQ-DI is derived from the HAQ, Health Assessment Questionnaire, developed in the 1980's. The HAQ-DI measures the quality of life of the patient by asking the patient to report answers to their abilities to perform daily life tasks such as getting in and out of bed. It ranges from 0 to a maximum value of 3. Values in the range of 0 to 1 implies the patient has mild difficulties to moderate disability, 1 to 2 implies that the patient has a moderate to severe disability, and 2 to 3 implies a very severe disability.
  units on a scale | 1.47 (0.60)
Max Joint Power Doppler Ultrasound (PDUS) [Mean (Standard Deviation); unit: units on a scale] — 34 joints will be evaluated using a 0 to 3 point scale for each joint and the sum of these represents PDUS. The Power Doppler Synovitis Score (PDUS) ranges from 0 to 102. Scores of 0 indicate the least amount of inflammation of the joint while scores of 3 indicate the most amount of inflammation. A higher value of the total score for PDUS represents more severe disease level.
  units on a scale | 29.59 (16.06)
Max Joint Grey-Scale Ultrasound (GSUS) [Mean (Standard Deviation); unit: units on a scale] — 34 joints will be evaluated using a 0 to 3 point scale for each joint and the sum of these represents GSUS. The grey scale synovial hypertrophy score (GSUS) ranges from 0 to 102. Scores of 0 indicate the least amount of inflammation of the joint while scores of 3 indicate the most amount of inflammation. A higher value of the total score for GSUS represents more severe disease level.
  units on a scale | 43.61 (14.68)

OUTCOME MEASURES:

1. Primary Outcome: Baseline to Month 3 Change in Total Power Doppler Synovitis Score of 34 Joints (Range 0 - 102)
Description: 34 joints will be evaluated using a 0 to 3 point scale for each joint. Power Doppler synovitis score is the sum of all the joint scores. Change scores are calculated by subtracting Baseline minus 3 Month Power Doppler scores.
  This scale is called the Power Doppler Synovitis Score (PDUS). It ranges from 0 to 102. Scores of 0 indicate the least amount of inflammation of the joint while scores of 3 indicate the most amount of inflammation. Therefore, a higher value of the total score for PDUS represents more severe disease level.
Time Frame: Baseline, 3 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Change of Total Power Doppler Synovitis Score 3 Month: All subjects will receive tocilizumab.
  Tocilizumab: All subjects will start at 4mg/kg. After 3 months, if DAS28 > 3.2, dosage will be escalated to 8 mg/kg.
Arm/Group | Mean Change of Total Power Doppler Synovitis Score 3 Month
Number analyzed (Participants) | 50
units on a scale | 6.84 (13.09)

2. Secondary Outcome: Baseline to Month 6 Change in Total Power Doppler Synovitis Score of 34 Joints (Range 0 - 102)
Description: 34 joints will be evaluated using a 0 to 3 point scale for each joint. Power Doppler synovitis score is the sum of all the joint scores. Change scores are calculated by subtracting Baseline minus 6 Month Power Doppler scores.
  This scale is called the Power Doppler Synovitis Score (PDUS). It ranges from 0 to 102. Scores of 0 indicate the least amount of inflammation of the joint while scores of 3 indicate the most amount of inflammation. Therefore, a higher value of the total score for PDUS represents more severe disease level.
Time Frame: Baseline, 6 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Change of Total Power Doppler Synovitis Score 6 Month: All subjects will receive tocilizumab.
  Tocilizumab: All subjects will start at 4mg/kg. After 3 months, if DAS28 > 3.2, dosage will be escalated to 8 mg/kg.
Arm/Group | Mean Change of Total Power Doppler Synovitis Score 6 Month
Number analyzed (Participants) | 44
units on a scale | 13.16 (15.68)

3. Secondary Outcome: Baseline to Month 3 Change in Total B-mode Synovial Hypertrophy Score of 34 Joints
Description: 34 joints will be evaluated using a 0 to 3 point scale for each joint. Synovial hypertrophy score is the sum of all the joint scores. Change scores are calculated by subtracting Baseline minus 3 Month Synovial Hypertrophy Scores.
  This scale is called the Grey Scale Synovial Hypertrophy Score (GSUS). Please note that B-mode is the same as GSUS. It ranges from 0 to 102. Scores of 0 indicate the least amount of inflammation of the joint while scores of 3 indicate the most amount of inflammation. Therefore, a higher value of the total score for GSUS represents more severe disease level.
Time Frame: Baseline, 3 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Change Total B-mode Synovial Hypertrophy Score 3 Month: All subjects will receive tocilizumab.
  Tocilizumab: All subjects will start at 4mg/kg. After 3 months, if DAS28 > 3.2, dosage will be escalated to 8 mg/kg.
Arm/Group | Mean Change Total B-mode Synovial Hypertrophy Score 3 Month
Number analyzed (Participants) | 50
units on a scale | 5.26 (12.55)

4. Secondary Outcome: Baseline to Month 6 Change in Total B-mode Synovial Hypertrophy Score of 34 Joints
Description: 34 joints will be evaluated using a 0 to 3 point scale for each joint. Synovial hypertrophy score is the sum of all the joint scores. Change scores are calculated by subtracting Baseline minus 6 Month Synovial Hypertrophy Scores.
  This scale is called the Grey Scale Synovial Hypertrophy Score (GSUS). Please note that B-mode is the same as GSUS. It ranges from 0 to 102. Scores of 0 indicate the least amount of inflammation of the joint while scores of 3 indicate the most amount of inflammation. Therefore, a higher value of the total score for GSUS represents more severe disease level.
Time Frame: Baseline, 6 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Change Total B-mode Synovial Hypertrophy Score 6 Month: All subjects will receive tocilizumab.
  Tocilizumab: All subjects will start at 4mg/kg. After 3 months, if DAS28 > 3.2, dosage will be escalated to 8 mg/kg.
Arm/Group | Mean Change Total B-mode Synovial Hypertrophy Score 6 Month
Number analyzed (Participants) | 44
units on a scale | 11.00 (15.32)

5. Secondary Outcome: Baseline to Month 3 Change in DAS28/ESR
Description: 28 joints will be evaluated for Tender Joint Count (TJC) and Swollen Joint Count (SJC) as well as patient and physician global values assessed at the time of each visit, finally the ESR lab value will be included in the total calculation. Change scores are calculated by subtracting Baseline minus 3 Month Disease Activity Score (DAS) scores.
  The scale being used is called the Disease Activity Score for 28 Joints (DAS28) using the Erythrocyte Sedimentation Rate (ESR) in the calculation rather than the C Reactive Protein (CRP). The scale ranges from 0 to 9.4. Values of DAS28 below 2.6 imply remission, below 3.2 imply low disease activity and greater than 5.1 implies active disease.
Time Frame: Baseline, 3 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Change in DAS28/ESR 3 Month: All subjects will receive tocilizumab.
  Tocilizumab: All subjects will start at 4mg/kg. After 3 months, if DAS28 > 3.2, dosage will be escalated to 8 mg/kg.
Arm/Group | Mean Change in DAS28/ESR 3 Month
Number analyzed (Participants) | 50
units on a scale | 1.20 (1.08)

6. Secondary Outcome: Baseline to Month 6 Change in DAS28/ESR
Description: 28 joints will be evaluated for TJC and SJC as well as patient and physician global values assessed at the time of each visit, finally the ESR lab value will be included in the total calculation. Change scores are calculated by subtracting Baseline minus 6 Month DAS scores.
  The scale being used is called the Disease Activity Score for 28 Joints (DAS28) using the Erythrocyte Sedimentation Rate (ESR) in the calculation rather than the C Reactive Protein (CRP). The scale ranges from 0 to 9.4. Values of DAS28 below 2.6 imply remission, below 3.2 imply low disease activity and greater than 5.1 implies active disease.
Time Frame: Baseline, 6 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Change in DAS28/ESR 6 Month: All subjects will receive tocilizumab.
  Tocilizumab: All subjects will start at 4mg/kg. After 3 months, if DAS28 > 3.2, dosage will be escalated to 8 mg/kg.
Arm/Group | Mean Change in DAS28/ESR 6 Month
Number analyzed (Participants) | 44
units on a scale | 2.32 (1.22)

7. Secondary Outcome: Baseline to Month 3 Change in CDAI
Description: 28 joints will be evaluated for TJC and SJC as well as patient and physician global values assessed at the time of each visit. Change scores are calculated by subtracting Baseline minus 3 Month CDAI scores.
  The scale being used is called the Clinical Disease Activity Index (CDAI) and has a range of 0 to 76. Values of CDAI below 2.8 imply remission, below 10 imply low disease activity, below 22 imply moderate disease activity, and above 22 implies high disease activity.
Time Frame: Baseline, 3 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Change in CDAI 3 Month: All subjects will receive tocilizumab.
  Tocilizumab: All subjects will start at 4mg/kg. After 3 months, if DAS28 > 3.2, dosage will be escalated to 8 mg/kg.
Arm/Group | Mean Change in CDAI 3 Month
Number analyzed (Participants) | 50
units on a scale | 9.64 (10.72)

8. Secondary Outcome: Baseline to Month 6 Change in CDAI
Description: 28 joints will be evaluated for TJC and SJC as well as patient and physician global values assessed at the time of each visit. Change scores are calculated by subtracting Baseline minus 6 Month CDAI scores.
  The scale being used is called the Clinical Disease Activity Index (CDAI) and has a range of 0 to 76. Values of CDAI below 2.8 imply remission, below 10 imply low disease activity, below 22 imply moderate disease activity, and above 22 implies high disease activity.
Time Frame: Baseline, 6 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Change in CDAI 6 Month: All subjects will receive tocilizumab.
  Tocilizumab: All subjects will start at 4mg/kg. After 3 months, if DAS28 > 3.2, dosage will be escalated to 8 mg/kg.
Arm/Group | Mean Change in CDAI 6 Month
Number analyzed (Participants) | 44
units on a scale | 16.70 (12.27)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Tocilizumab
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 1/54
Other Adverse Events (participants affected / at risk) | 51/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=54)
Breast Cancer (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=54)
Abdominal Pain (Gastrointestinal disorders) | 3
Anemia (Blood and lymphatic system disorders) | 5
Bruises on Different Body Sites (Vascular disorders) | 6
Diarrhea (Gastrointestinal disorders) | 6
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyslipidemia (Blood and lymphatic system disorders) | 3
Falling Down (General disorders) | 3
Fatigue (General disorders) | 4
Headaches (General disorders) | 10
Hypercholesterolemia (Cardiac disorders) | 17
Hypertension (Vascular disorders) | 3
Hypokalemia (Blood and lymphatic system disorders) | 8
Increased Pain (General disorders) | 3
Insomnia (General disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 12
Loose Stool (Gastrointestinal disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 4
Rheumatoid Arthritis Flare (Musculoskeletal and connective tissue disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 21
Urinary Tract Infection (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT01717859/Prot_SAP_000.pdf